CLINICAL TRIAL: NCT01392807
Title: An Open-label, Single-center Study to Assess the Pharmacokinetics of NKTR-118 in Patients With Impaired Hepatic Function and Subjects With Normal Hepatic Function Following Administration of a Single Dose of 25mg NKTR-118
Brief Title: Open-label Study to Assess the Pharmacokinetics of NKTR-118 in Patients With Impaired Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: D3820C00010
Record Dates: First submitted 2011-07-08; First posted 2011-07-13 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Hepatic; Functional Disturbance
Keywords: Phase 1; volunteers with hepatic impairment; pharmacokinetics; NKTR-118; Child-Pugh scale; AUC; Cmax; tmax; t1/2
MeSH Terms: interventions — naloxegol

ARMS (3):
- Group 1 (Experimental): Normal hepatic function, 25 mg NKTR-118 administered orally
  Interventions: Drug: NKTR-118
- Group 2 (Experimental): Mild hepatic impairment, 25 mg NKTR-118 administered orally
  Interventions: Drug: NKTR-118
- Group 3 (Experimental): Moderate hepatic impairment, 25 mg NKTR-118 administered orally
  Interventions: Drug: NKTR-118

INTERVENTIONS:
Drug: NKTR-118 — 25 mg Oral tablets, single dose

SUMMARY:
The purpose of this study is to assess the pharmacokinetics of NKTR-118 in patients with impaired hepatic function versus subjects with normal hepatic function.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged 18 years or more with a weight of at least 50 kg and BMI between 18 and 40 kg/m2, inclusive.
* Negative screen for human immunodeficiency virus (HIV)
* For subjects with normal hepatic function, negative results for serum hepatitis B (HBV) surface antigen, HCV antibody, and HIV

Exclusion Criteria:

* Plasma or blood product donation within 1 month of screening or any blood donation/blood loss greater than 500 mL during the 3 months prior to screening.
* History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity
* Known or suspected history of drug/chemical abuse within the past 2 years as judged by the Investigator.
* Subjects with a history of surgery on the gastrointestinal tract.
* For patients with hepatic impairment, fluctuating or rapidly deteriorating hepatic function as indicated by clinical and/or laboratory signs of hepatic impairment (e.g. advanced ascites, infection of ascites, fever, or active gastrointestinal bleeding).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-07; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
To assess the pharmacokinetics of a single dose of NKTR-118 25 mg by assessment of area under the curve over the time (AUC) and maximum concentration (Cmax) | Duration from predose day 1 to day 6.

SECONDARY OUTCOMES:
To examine the safety and tolerability of a single oral dose of 25 mg NKTR-118 in patients with impaired hepatic function and in subjects with normal hepatic function by collecting adverse events. | Duration from day -1 to follow up. ( Approximately 15-18 days)
To examine the safety and tolerability of a single oral dose of 25 mg NKTR-118 in patients with impaired hepatic function and in subjects with normal hepatic function by collecting vital signs | Duration from day -1 to follow up. ( Approximately 15-18 days)
To examine the safety and tolerability of a single oral dose of 25 mg NKTR-118 in patients with impaired hepatic function by collecting safety blood samples | Duration from day -1 to follow up. ( Approximately 15-18 days)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Sostek, MD, Study Director — AstraZeneca; Thomas Marbury, MD, Principal Investigator — Orlando Clinical Research Center; Bo Fransson, MD, Study Chair — AstraZeneca
Locations (1):
- Research Site, Overland Park, Kansas, United States

REFERENCES:
- [Derived] Bui K, She F, Sostek M. The effects of mild or moderate hepatic impairment on the pharmacokinetics, safety, and tolerability of naloxegol. J Clin Pharmacol. 2014 Dec;54(12):1368-74. doi: 10.1002/jcph.348. Epub 2014 Jun 27. PMID 24945932
- See also: D3820C00010 Clinical Study Report Synopsis.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1392&filename=D3820C00010_Clinical_Study_Report_Synopsis.pdf